CLINICAL TRIAL: NCT04717661
Title: A Diagnostic Test Study of Characteristic Sound Waves in Radial Artery of Early Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Qianfoshan Hospital (Other)
Responsible Party: Principal Investigator, Lili Cao, dean of orthopedic department, Qianfoshan Hospital
Other Study IDs: SFUYIN-01
Record Dates: First submitted 2021-01-18; First posted 2021-01-22 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-01

CONDITIONS: Early Pregnancy; Radial Artery
Keywords: Early Pregnancy; Diagnostic Test; Radial Artery; Sound Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 76 healthy early pregnant women in the trial group: The pulse sound waves of three parts and five layers of each of the two hands of 76 pregnant women will be collected by Pulse Detection System of Sound Waves.
- 76 relatively healthy non-pregnant women in the control group: The pulse sound waves of three parts and five layers of each of the two hands of 76 relatively healthy non-pregnant women will be collected by Pulse Detection System of Sound Waves.

SUMMARY:
Pulse diagnosis is an important method to judge the status of patients in the process of diagnosis and treatment of traditional Chinese medicine. At present, the commonly used site of pulse diagnosis is the radial artery, which is divided into "cun""guan""chi". Whether the diagnosis of pregnancy can be diagnosed by pulse diagnosis has been perplexing clinicians. In long-term clinical practice, it is found that slippery pulse often occurs in the radial artery of pregnant women. Before the 13th week of pregnancy, it is called early pregnancy. During pregnancy, chorionic gonadotropin gradually increases, progesterone increases, humoral metabolism changes, blood volume increases, hemodilution and cardiac output increase. Other studies have shown that due to the effect of estrogen, the number of active levels of renin in plasma increase several times, and will increase with the progression of pregnancy. This series of changes in pregnant women may be reflected in the pulse. During the clinical pulse examination, our team has found that some pregnant women had no abnormality in pre-pregnancy examination such as B-ultrasound, and abnormal unsmooth pulse in the ulna could be felt during pulse examination. Through follow-up, it is found that this kind of pregnant women may have miscarriage or stillbirth.

Our team found that there are low-frequency sound waves in the radial artery, which carry the physiological and pathological information of the organs in the body, and developed a "Pulse Detection System of Sound Waves". Previous projects have explored the abnormal sound waves of radial artery in patients with sequelae of cerebral infarction, stable coronary heart disease, chronic gastritis, neck-shoulder syndrome, liver cirrhosis and other diseases and achieved certain results.

Therefore, in this study, the "Pulse Detection System of Sound Waves" will be used to collect the sound waves in the radial artery of 76 healthy early pregnant women and 76 relatively healthy non-pregnant women. Fourier transform, wavelet analysis, Hilbert yellow transform and other methods will be used to identify the different characteristics of the pulse acoustic signals, and observe the time-frequency domain characteristics of the trial group and the control group.And researchers will carry on the diagnostic test, calculate the sensitivity and specificity of the "Pulse Detection System of Sound Waves" in the diagnosis of pregnancy. This study will verify the efficacy of pulse diagnosis of traditional Chinese medicine in the diagnosis of pregnancy and lay a foundation for the diagnosis of abnormal pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Trial group:

1. Pregnant women who have been diagnosed as early pregnancy by laboratory and ultrasound;
2. First-born singleton pregnancy, from 6 weeks to 13 weeks;
3. There are no pregnancy complications, the vital signs were stable, and the results of biochemical tests were normal;
4. Patients with informed consent to accept this pulse collection.

Control group:

1. The inclusion of relatively healthy women is those with negative diagnostic criteria for early pregnancy pregnant women;
2. Patients with informed consent to accept this pulse collection;
3. The vital signs were stable, the results of biochemical tests were normal, and there were no severe diseases of brain, liver and kidney.

Exclusion Criteria:

Trial group:

1. Pregnant women with ovarian, fallopian tube, uterine diseases, hypertension and diabetes during pregnancy;
2. Definitely diagnose patients with respiratory, cardiovascular, cerebrovascular, liver and kidney, blood, endocrine and other system diseases and severe infectious diseases;
3. Those who have had a cesarean section; history of miscarriage；
4. Those who have a severe illness and sit for less than 10 minutes in a quiet state;
5. Patients with mental illness, depression, and cognitive impairment;
6. Pulse on back of wrist, oblique-running pulse, etc. who are not easy to collect pulse;
7. Those who have incomplete information due to subjective or objective reasons that affect the result judgment;
8. Patients with Parkinson's or other limb tremors;

Control group:

1. Those who have had a history of miscarriage or ectopic pregnancy;
2. Patients with severe infectious diseases;
3. Pulse on back of wrist, oblique-running pulse, etc. who are not easy to collect pulse;
4. The incomplete information affects the judgment of the result due to subjective or objective reasons;
5. Patients with Parkinson's or other limb tremors;
6. Menstrual women.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Early pregnancy women and relatively healthy non-pregnant women.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-03-01 (Estimated)

PRIMARY OUTCOMES:
Frequencies of characteristic sound waves in the pulses | The data will be collected,analyzed and calculated in about 7 days.
  Using Pulse Detection System of Sound Waves (PDSSW) to collect the pulse waves of both hands.The percentage(%) of frequencies of characteristics sound waves in the pulse will be calculated.
The changes of sound waves in the pulses | The discovery of characteristic sound waves may take three months.
  The changes of sound waves in the early pregnant women at different hertz(Hz) frequencies and SMPL amplitudes will be compared with relatively healthy women's.
Diagnostic test | Diagnostic tests may take about 1 month.
  The percentage(%) of sensitivity,specificity positive likelihood ratio and negative likelihood ratio of the ''Pulse Detection System of Sound Waves'' in the diagnosis of early pregnant women.
Sound waves analysis | 1 month
  The Hertz(Hz) of the different segments of sound waves in Wavelet transform; The Hertz(Hz) of the different layers of the sound waves in Hilbert-Huang;The SMPL amplitudes of sound waves in Discrete Fourier Transform;The sample Entropy(sampEn) of sound waves in Sample Entropy.
  time-frequency characteristics, time-domain characteristics and frequency-domain features will be extracted.

CONTACTS AND LOCATIONS:
Overall Officials: Lucheng Song, Doctor, Principal Investigator — The First Affiliated Hospital of Shandong First Medical University & Shandong Provincial Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, The First Hospital affiliated of Shandong First Medical University, Jinan, Shandong, China

REFERENCES:
- [Background] Carusi D. Pregnancy of unknown location: Evaluation and management. Semin Perinatol. 2019 Mar;43(2):95-100. doi: 10.1053/j.semperi.2018.12.006. Epub 2018 Dec 20. PMID 30606496
- [Background] Drukker L, Droste R, Chatelain P, Noble JA, Papageorghiou AT. Safety Indices of Ultrasound: Adherence to Recommendations and Awareness During Routine Obstetric Ultrasound Scanning. Ultraschall Med. 2020 Apr;41(2):138-145. doi: 10.1055/a-1074-0722. Epub 2020 Feb 27. PMID 32107757
- [Background] Bilton K, Hammer L, Zaslawski C. Contemporary Chinese pulse diagnosis: a modern interpretation of an ancient and traditional method. J Acupunct Meridian Stud. 2013 Oct;6(5):227-33. doi: 10.1016/j.jams.2013.04.002. Epub 2013 Apr 24. PMID 24139459
- [Background] Lumbers ER, Pringle KG. Roles of the circulating renin-angiotensin-aldosterone system in human pregnancy. Am J Physiol Regul Integr Comp Physiol. 2014 Jan 15;306(2):R91-101. doi: 10.1152/ajpregu.00034.2013. Epub 2013 Oct 2. PMID 24089380
- [Background] Tkachenko O, Shchekochikhin D, Schrier RW. Hormones and hemodynamics in pregnancy. Int J Endocrinol Metab. 2014 Apr 1;12(2):e14098. doi: 10.5812/ijem.14098. eCollection 2014 Apr. PMID 24803942
- [Background] Rodger M, Sheppard D, Gandara E, Tinmouth A. Haematological problems in obstetrics. Best Pract Res Clin Obstet Gynaecol. 2015 Jul;29(5):671-84. doi: 10.1016/j.bpobgyn.2015.02.004. Epub 2015 Mar 4. PMID 25819750
- [Background] Li K, Zhang S, Yang L, Jiang H, Chi Z, Wang A, Yang Y, Li X, Hao D, Zhang L, Zheng D. Changes of Arterial Pulse Waveform Characteristics with Gestational Age during Normal Pregnancy. Sci Rep. 2018 Oct 22;8(1):15571. doi: 10.1038/s41598-018-33890-1. PMID 30349022
- [Background] Li K, Zhang S, Chi Z, Yang Y, Jiang H, Yang L, Wang A, Zhang L, Chen F, Zheng D. Arterial Pulse Waveform Characteristics Difference between the Three Trimesters of Healthy Pregnant Women. Annu Int Conf IEEE Eng Med Biol Soc. 2018 Jul;2018:5317-5320. doi: 10.1109/EMBC.2018.8513492. PMID 30441537